CLINICAL TRIAL: NCT02800356
Title: Subthreshold Laser Treatment for Reticular Pseudodrusen and Incipient Geographic Atrophy Secondary to Age - Related Macular Degeneration: a Pilot Study
Brief Title: Subthreshold Laser Treatment for Reticular Pseudodrusen and Geographic Atrophy Secondary to AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Querques Giuseppe, Head-Medical retina & Imaging unit, Ospedale San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PASCAL-GA
Record Dates: First submitted 2016-06-02; First posted 2016-06-15 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Age-Related Macular Degeneration; Geographic Atrophy; Reticular Pseudodrusen
Keywords: Age-Related Macular Degeneration; Geographic Atrophy; Reticular pseudodrusen; Lasers; PASCAL 577
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pseudodrusen (Experimental): Subthreshold 577 nm yellow wavelength laser photo-coagulator
  Interventions: Procedure: Subthreshold 577 nm yellow wavelength laser photo-coagulator
- Geographic atrophy (Experimental): Subthreshold 577 nm yellow wavelength laser photo-coagulator
  Interventions: Procedure: Subthreshold 577 nm yellow wavelength laser photo-coagulator

INTERVENTIONS:
Procedure: Subthreshold 577 nm yellow wavelength laser photo-coagulator — Subthreshold photocoagulation is a method in which the burn spots (treated areas) cannot be seen with biomicroscopy, on color fundus photograph, on Optical Coherence Tomography or Fluorescein Angiography when the subthreshold level is adequately set. Subthreshold photocoagulation can be considered to be truly minimally invasive or non-damaging photocoagulation. A term sometimes used is photo-thermal stimulation since the Retinal Pigment Epithelium (RPE) layer is heated and stimulated, but not destroyed.
  The threshold level output power is set to obtain barely visible burn at approximately 200 mW to 250 mW using the titration mode, and irradiation is conducted after switching over to Endpoint Management.
  Other Names: Pascal Synthesis 577 (Topcon); Subthreshold laser

SUMMARY:
To evaluate the effectiveness of subthreshold laser treatment on retinal sensitivity in patients with reticular pseudodrusen and incipient Geographic Atrophy (GA) secondary to Age-Related Macular Degeneration (AMD). Secondary objective is to investigate changes in best-corrected visual acuity, atrophy progression and safety.

ELIGIBILITY:
Inclusion Criteria:

* GA < 0.5 disk areas secondary to AMD and/or Reticular pseudodrusen
* 50 years or older
* The periphery of the atrophic lesions must demonstrate increased autofluorescence
* Best corrected visual acuity between 20/20 and 20/400 inclusive
* Clear ocular media
* Ability to provide informed consent and attend all study visits

Exclusion Criteria:

* GA secondary to other causes aside from AMD
* Evidence of choroidal neovascularization in either eye
* Any prior treatment for AMD, aside from antioxidants
* Any other ocular condition that would progress in the study period and confound visual acuity assessment
* Any ocular or systemic medication known to be toxic to the lens, retina or optic nerve
* Presence of idiopathic or autoimmune-associated uveitis
* Any intraocular surgery 3 months of entry
* Any prior thermal laser in the macula
* History of vitrectomy, filtering surgery, corneal transplant or retinal detachment surgery
* Previous therapeutic radiation in the ocular region in either eye
* Any treatment with an investigational agent in the previous 60 days before study entry
* Women of child-bearing potential, defined as all women less than 1 year postmenopausal or less than 6 weeks since sterilization at Baseline, unless they are using highly effective methods of contraception during dosing of study treatment
* Participation in an investigational drug, biologic, or device study within 6 Months prior to Baseline [Note: observational clinical studies solely involving over-the-counter vitamins, supplements, or diets are not exclusionary

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Querques, MD, PhD, Principal Investigator — Ospedale San Raffaele; Riccardo Sacconi, MD, Principal Investigator — Ospedale San Raffaele; Francesco Gelormini, MDs, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luttrull JK, Musch DC, Mainster MA. Subthreshold diode micropulse photocoagulation for the treatment of clinically significant diabetic macular oedema. Br J Ophthalmol. 2005 Jan;89(1):74-80. doi: 10.1136/bjo.2004.051540. PMID 15615751
- [Background] Parodi MB, Spasse S, Iacono P, Di Stefano G, Canziani T, Ravalico G. Subthreshold grid laser treatment of macular edema secondary to branch retinal vein occlusion with micropulse infrared (810 nanometer) diode laser. Ophthalmology. 2006 Dec;113(12):2237-42. doi: 10.1016/j.ophtha.2006.05.056. Epub 2006 Sep 25. PMID 16996596
- [Background] Chen SN, Hwang JF, Tseng LF, Lin CJ. Subthreshold diode micropulse photocoagulation for the treatment of chronic central serous chorioretinopathy with juxtafoveal leakage. Ophthalmology. 2008 Dec;115(12):2229-34. doi: 10.1016/j.ophtha.2008.08.026. PMID 19041477
- [Background] Luttrull JK, Sinclair SH. Safety of transfoveal subthreshold diode micropulse laser for fovea-involving diabetic macular edema in eyes with good visual acuity. Retina. 2014 Oct;34(10):2010-20. doi: 10.1097/IAE.0000000000000177. PMID 24837050
- [Background] Luttrull JK, Chang DB, Margolis BW, Dorin G, Luttrull DK. LASER RESENSITIZATION OF MEDICALLY UNRESPONSIVE NEOVASCULAR AGE-RELATED MACULAR DEGENERATION: Efficacy and Implications. Retina. 2015 Jun;35(6):1184-94. doi: 10.1097/IAE.0000000000000458. PMID 25650711
- [Background] Vujosevic S, Martini F, Longhin E, Convento E, Cavarzeran F, Midena E. SUBTHRESHOLD MICROPULSE YELLOW LASER VERSUS SUBTHRESHOLD MICROPULSE INFRARED LASER IN CENTER-INVOLVING DIABETIC MACULAR EDEMA: Morphologic and Functional Safety. Retina. 2015 Aug;35(8):1594-603. doi: 10.1097/IAE.0000000000000521. PMID 25719988
- [Background] Bessho K, Rodanant N, Bartsch DU, Cheng L, Koh HJ, Freeman WR. Effect of subthreshold infrared laser treatment for drusen regression on macular autofluorescence in patients with age-related macular degeneration. Retina. 2005 Dec;25(8):981-8. doi: 10.1097/00006982-200512000-00005. PMID 16340527
- [Background] Virgili G, Michelessi M, Parodi MB, Bacherini D, Evans JR. Laser treatment of drusen to prevent progression to advanced age-related macular degeneration. Cochrane Database Syst Rev. 2015 Oct 23;2015(10):CD006537. doi: 10.1002/14651858.CD006537.pub3. PMID 26493180

RESULTS

PARTICIPANT FLOW:
Groups:
- Pseudodrusen: Patients affected by reticular pseudodrusen secondary to AMD were included and treated by subthreshold 577 nm yellow wavelength laser photo-coagulator.
Period: Overall Study
Arm/Group | Pseudodrusen
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pseudodrusen
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 20
Retinal sensitivity in the treated area [Mean (Standard Deviation); unit: dB] | 12.08 (4.65)

OUTCOME MEASURES:

1. Primary Outcome: Retinal Sensitivity
Description: Change in retinal sensitivity on customized microperimetry (treated area).
Time Frame: Baseline, 4 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Pseudodrusen
Number analyzed (Participants) | 20
dB
  Baseline | 12.08 (4.65)
  4 weeks | 11.08 (5.06)
  12 weeks | 11.45 (5.70)
Statistical Analysis 1: Comparison: Pseudodrusen; Test type: Other; p = 0.404, ANOVA; Analysis of Variance (ANOVA) for paired samples with Bonferroni post-hoc analysis

2. Secondary Outcome: Visual Acuity
Description: Change in mean Visual Acuity
Time Frame: Baseline, 4 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Pseudodrusen
Number analyzed (Participants) | 20
LogMAR
  Baseline | 0.14 (0.09)
  4 weeks | 0.135 (0.10)
  12 weeks | 0.115 (0.09)
Statistical Analysis 1: Comparison: Pseudodrusen; Test type: Other; p = 0.232, ANOVA; Analysis of Variance (ANOVA) for paired samples with Bonferroni post-hoc analysis

3. Secondary Outcome: The Thickness of the Outer Nuclear Layer in the Treated Area
Description: The thickness of the outer nuclear layer in the treated area was measured using structural OCT
Time Frame: Baseline, 4 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Pseudodrusen
Number analyzed (Participants) | 20
µm
  Baseline | 59.30 (13.50)
  4 weeks | 64.75 (12.31)
  12 weeks | 67.75 (15.52)
Statistical Analysis 1: Comparison: Pseudodrusen; Test type: Other; p = 0.001, ANOVA; Analysis of Variance (ANOVA) for paired samples with Bonferroni post-hoc analysis

4. Secondary Outcome: Number of Partecipants With Adverse and Serious Adverse Events
Description: Adverse and Serious Adverse Events were recorded
Time Frame: 4 weeks and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pseudodrusen
Number analyzed (Participants) | 20
Participants | 0

5. Secondary Outcome: Number of Partecipants With Presence of Haemorrhage, Photocoagulation Spots, Ischemic Areas
Description: Fundus examination by using slit-lamp was performed in order to assess the presence of hemorrhage, photocoagulation spots, ischemic areas
Time Frame: 4 weeks and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pseudodrusen
Number analyzed (Participants) | 20
Participants | 0

6. Secondary Outcome: Intraocular Pressure
Description: Intraocular pressure was recorded.
Time Frame: 4 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pseudodrusen
Number analyzed (Participants) | 20
mmHg
  Baseline | 15.5 (2.9)
  4 weeks | 14.9 (2.4)
  12 weeks | 14.7 (2.4)
Statistical Analysis 1: Comparison: Pseudodrusen; Test type: Other; p = 0.267, ANOVA; Analysis of Variance (ANOVA) for paired samples with Bonferroni post-hoc analysis

ADVERSE EVENTS:
Time Frame: 12 weeks.
Arm/Group | Pseudodrusen
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT02800356/Prot_SAP_000.pdf